CLINICAL TRIAL: NCT04070560
Title: SAVE (Sustained Cord Circulation Awaiting VEntilation)
Brief Title: Effects of Delayed Cord Clamping During Resuscitation of Newborn Near Term and Term Infants
Acronym: SAVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAVE1
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Asphyxia Neonatorum; Resuscitation
Keywords: umbilical cord
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Resuscitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early (≤ 60 seconds) cord clamping (Active Comparator): If the infant don't breathe, the umbilical cord is clamped (≤ 60 seconds) and cut and resuscitation will be provided at a resuscitation table Other Name: Immediate clamping
  Interventions: Procedure: Early (≤ 60 seconds) cord clamping
- Intact cord (≥ 180 seconds) resuscitation (Active Comparator): If the infant don't breathe, the umbilical cord is not clamped and cut until after 180 seconds. Initial resuscitation will be provided bedside to the mother
  Other Names:
  Late cord clamping Deferred cord clamping Optimal cord clamping
  Interventions: Procedure: Intact cord (≥ 180 seconds) resuscitation

INTERVENTIONS:
Procedure: Intact cord (≥ 180 seconds) resuscitation — Resuscitation performed in near proximity to the mother with umbilical cord uncut
  Arms: Intact cord (≥ 180 seconds) resuscitation
Procedure: Early (≤ 60 seconds) cord clamping — Resuscitation performed at a designated area after umbilical cord is cut
  Arms: Early (≤ 60 seconds) cord clamping

SUMMARY:
This study evaluates resuscitation with an intact umbilical cord compared to resuscitation with the umbilical cord cut. Half of the newborn babies in need of resuscitation will be handled while having an intact umbilical cord and half will have their umbilical cord cut.

DETAILED DESCRIPTION:
The routine procedure when a newborn baby is in need of resuscitation is to cut the umbilical cord and move the baby to a designated area for resuscitation, which can include stimulation, clearing the airways, administration of oxygen and/or positive pressure ventilation by bag and mask och T-piece resuscitator.

It has been suggested, and pilot studies has shown preliminary results, that keeping the umbilical cord intact while performing resuscitation may improve the babies outcome, by continued exchange of oxygen and carbon dioxide be the placenta and facilitating the neonatal pulmonary and circulatory transition.

Because of the limiting length of the umbilical cord, resuscitation with an intact cord must be performed in close proximity to the mother.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy week ≥35 + 0
* Singletons
* Expected vaginal delivery
* The woman / couple can adequately assimilate information about the study
* Signed informed consent of both prospective parents

Exclusion Criteria:

* Congenital malformation that complicates resuscitation (such as severe malformation of mouth, pharynx, respiratory system) or which causes the child not to be resuscitated due to internal structural malformations (such as more severe heart failure, diaphragm fractures, etc.)
* The child is born via acute caesarean section after inclusion and opening of study envelope
* placenta abruption / or damage to umbilical cord during childbirth (when circulation through an intact umbilical cord cannot be achieved after birth)

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Apgar score | At 5 minutes after birth
  Assessed by staff, composite of heart rate, breathing effort, skin color, muscle tone and reflexes, each sub scale 0 (absent), 1, 2 (normal). Minimum 0, maximum 10. Less than 4 is a measure for severe asphyxia, less than 7 measure of mild asphyxia.

SECONDARY OUTCOMES:
Apgar score | At 1 minute after birth
  Assessed by staff, composite of heart rate, breathing effort, skin color, muscle tone and reflexes, each sub scale 0 (absent), 1, 2 (normal). Minimum 0, maximum 10. Less than 4 is a measure for severe asphyxia, less than 7 measure of mild asphyxia.
Apgar score | At 10 minute after birth
  Assessed by staff, composite of heart rate, breathing effort, skin color, muscle tone and reflexes, each sub scale 0 (absent), 1, 2 (normal). Minimum 0, maximum 10. Less than 4 is a measure for severe asphyxia, less than 7 measure of mild asphyxia.
Time of first cry or breathing effort | Within 10 minutes after birth
  Assessed by staff present
Time of establishing spontaneous breathing | Within 10 minutes after birth
  Assessed by staff present
Presence at one day of age | 24 hours
  The place of stay for newborn at one day of age
Need of neonatal intensive care | 7 days
  Admission to neonatal intensive care unit
Score for Neonatal Acute Physiology (SNAP-II) | 7 days
  Assessed by staff at neonatal intensive care unit
Morbidity Assessment Index for Newborns (MAIN) | 7 days
  Assessed by staff at neonatal intensive care unit
Blood glucose | 4 hours after birth
  Sampled by staff at nursery of neonatal intensive care
Breathing difficulties | 1 hours after birth
  Respiratory rate > 60, grunting/shallow breathing, nostril flaring, retractions between or under the ribs) Assessed by staff at nursery of neonatal intensive care
Breathing difficulties | 6 hours after birth
  Respiratory rate > 60, grunting/shallow breathing, nostril flaring, retractions between or under the ribs) Assessed by staff at nursery of neonatal intensive care
Mortality | One year
  Death after birth
Development | 12 months
  Assessed by Ages and Stages Questionnaire (ASQ). Minimum 0, maximum 300. Consist of 30 questions answered Yes (10), Sometimes (5), Not Yet (0). Five sub scales with six questions each: Communication, Fine motor, Gross motor, Problem solving and Personal-Social. Worse outcome is considered mean minus 2 standard deviations.
Development | 24 months
  Neurocognitive assessment by Bayley-III (alternative Bayley-IV if available). Derives a developmental quotient (DQ) three main subtests; the Cognitive Scale, the Language Scale, and the Motor Scale. Is assessed by special staff and have standardized interpretations of results.
Autism | 24 months
  Screening by Modified Checklist for Autism in Toddlers (M-CHAT). 20-question test. Answers "yes" or "no". A total score of 2 and below on the first part of the M-CHAT indicate low autism risk, a total score of 3-7 indicates medium risk and prompts administration of the follow-up form. A total score of 8 or higher indicates high autism risk.
Development | 54 months
  Neurocognitive assessment by Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV). 14 subtests. The core subtests are required for the computation of the Verbal, Performance, and Full Scale intelligence quotient (IQ). Also, two other composites Processing Speed Quotient and General Language Composite.
  Quotient and Composite scores have a mean of 100 and a standard deviation of 15. Subtest scaled scores have a mean of 10 and a standard deviation of 3. For Quotient and Composite score:
  below 70 is Extremely Low, 70-79 is Borderline, 80-89 is Low Average, 90-109 is Average, 110-119 is High Average, 120-129 is Superior, 130+ is Very Superior.
Motor development | 54 months
  Assessed by Movement Assessment Battery for Children (ABC). The test contains 8 tasks covering the following 3 areas: Manual Dexterity, Ball Skills, Static and Dynamic Balance. Standard scores for each domain can be compared to normative data and interpreted in terms of percentile equivalents (a) ≤5th percentile reflecting definite motor impairment, (b) ≤15th percentile reflecting borderline motor impairment, or (c) >15th percentile reflecting no motor impairment.

OTHER OUTCOMES:
Thompson score | 1 hour after birth
  Assessed by staff at neonatal intensive care unit. A scoring system for hypoxic ischaemic encephalopathy in predicting neurodevelopmental outcome. Minimum 0 (normal), maximum 22. A score ≥12 is associated with adverse outcomes.
Thompson score | 6 hours after birth
  Assessed by staff at neonatal intensive care unit. A scoring system for hypoxic ischaemic encephalopathy in predicting neurodevelopmental outcome. Minimum 0 (normal), maximum 22. A score ≥12 is associated with adverse outcomes.
Thompson score | 12 hours after birth
  Assessed by staff at neonatal intensive care unit. A scoring system for hypoxic ischaemic encephalopathy in predicting neurodevelopmental outcome. Minimum 0 (normal), maximum 22. A score ≥12 is associated with adverse outcomes.
Thompson score | 24 hours after birth
  Assessed by staff at neonatal intensive care unit. A scoring system for hypoxic ischaemic encephalopathy in predicting neurodevelopmental outcome. Minimum 0 (normal), maximum 22. A score ≥12 is associated with adverse outcomes.
Thompson score | 48 hours after birth
  Assessed by staff at neonatal intensive care unit. A scoring system for hypoxic ischaemic encephalopathy in predicting neurodevelopmental outcome. Minimum 0 (normal), maximum 22. A score ≥12 is associated with adverse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Andersson, MD PhD, Principal Investigator — Lunds University/Skåne University Hospital
Locations (3):
- Sweden (3):
  - Hospital of Halland, Halmstad, Halland County
  - Skåne University Hospital, Malmo, Skåne County
  - Ystad hospital, Ystad

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal, and that most preferably have an approval from an independent review committee.

REFERENCES:
- [Background] Niermeyer S, Velaphi S. Promoting physiologic transition at birth: re-examining resuscitation and the timing of cord clamping. Semin Fetal Neonatal Med. 2013 Dec;18(6):385-92. doi: 10.1016/j.siny.2013.08.008. Epub 2013 Sep 19. PMID 24055300
- [Background] Katheria AC, Brown MK, Faksh A, Hassen KO, Rich W, Lazarus D, Steen J, Daneshmand SS, Finer NN. Delayed Cord Clamping in Newborns Born at Term at Risk for Resuscitation: A Feasibility Randomized Clinical Trial. J Pediatr. 2017 Aug;187:313-317.e1. doi: 10.1016/j.jpeds.2017.04.033. Epub 2017 May 16. PMID 28526223
- [Background] Katheria AC. Neonatal Resuscitation with an Intact Cord: Current and Ongoing Trials. Children (Basel). 2019 Apr 22;6(4):60. doi: 10.3390/children6040060. PMID 31013574
- [Background] Andersson O, Rana N, Ewald U, Malqvist M, Stripple G, Basnet O, Subedi K, Kc A. Intact cord resuscitation versus early cord clamping in the treatment of depressed newborn infants during the first 10 minutes of birth (Nepcord III) - a randomized clinical trial. Matern Health Neonatol Perinatol. 2019 Aug 29;5:15. doi: 10.1186/s40748-019-0110-z. eCollection 2019. PMID 31485335
- [Background] Ekelof K, Saether E, Santesson A, Wilander M, Patriksson K, Hesselman S, Thies-Lagergren L, Rabe H, Andersson O. A hybrid type I, multi-center randomized controlled trial to study the implementation of a method for Sustained cord circulation And VEntilation (the SAVE-method) of late preterm and term neonates: a study protocol. BMC Pregnancy Childbirth. 2022 Jul 26;22(1):593. doi: 10.1186/s12884-022-04915-5. PMID 35883044
- [Background] Wilander M, Sandblom J, Thies-Lagergren L, Andersson O, Svedenkrans J. Bilirubin Levels in Neonates >/=35 Weeks of Gestation Receiving Delayed Cord Clamping for an Extended Time-An Observational Study. J Pediatr. 2023 Jun;257:113326. doi: 10.1016/j.jpeds.2023.01.005. Epub 2023 Jan 14. PMID 36646247